CLINICAL TRIAL: NCT03302741
Title: Imaging of 3D Innervation Zone Distribution in Spastic Muscles From High-density Surface
Brief Title: Imaging of 3D Innervation Zone Distribution in Spastic Muscles From High-density Surface EMG Recordings
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: University of Houston (Other)
Responsible Party: Principal Investigator, Sheng Li, Professor, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-17-0174
Record Dates: First submitted 2017-10-01; First posted 2017-10-05 (Actual); Results first posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-10

CONDITIONS: Spasticity
Keywords: stroke
MeSH Terms: conditions — Muscle Spasticity; Stroke | interventions — Botulinum Toxins; Botulinum Toxins, Type A; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard BTX injection (ultrasound guided) (Active Comparator): For standard injection procedures, target muscles will be visualized under ultrasound imaging which is operated by an experienced and dedicated technician. Position of needle tip within the target muscle is visualized prior to injection. Ultrasound guidance can help ensure depth of needle tip location, i.e., to make sure the needle tip is within the muscle, but it is not able to tell where it is located with reference to the IZs of the entire muscle.
  Interventions: Drug: Botulinum neurotoxin (BTX); Other: Physical Therapy; Device: Standard BTX injection (ultrasound guided)
- 3-dimensional innervation zone (3DIZ) guided injection (Experimental): In the IZ-guided injection technique, IZ location obtained using the 3DIZ will be first marked over the skin surface of the muscle and the depth of the IZ will be also provided. The 3DIZ will be applied to the IZ-guided injection group 1 day prior to scheduled injection. The surface location and depth information of the IZ will be used to guide where the needle tip needs to go. Currently, patients commonly receive 1 to 2 injection sites, occasionally 3 sites for biceps muscles. To standardize the procedure, we will choose 2 sites for all patients.
  Interventions: Drug: Botulinum neurotoxin (BTX); Other: Physical Therapy; Device: 3-dimensional innervation zone (3DIZ) guided injection

INTERVENTIONS:
Drug: Botulinum neurotoxin (BTX) — Each patient will receive BTX injections in 2 sites. 100 units at double dilution will be injected at each site.
  Other Names: Botox
Other: Physical Therapy — Standard physical therapy will be ordered to both groups as part of standard of care for patients after BTX injections to maximize the outcomes.
Device: Standard BTX injection (ultrasound guided) — For standard injection procedures, target muscles will be visualized under ultrasound imaging which is operated by an experienced and dedicated technician. Position of needle tip within the target muscle is visualized prior to injection. Ultrasound guidance can help ensure depth of needle tip location, i.e., to make sure the needle tip is within the muscle, but it is not able to tell where it is located with reference to the innervation zones (IZs) of the entire muscle.
  Arms: Standard BTX injection (ultrasound guided)
Device: 3-dimensional innervation zone (3DIZ) guided injection — Simultaneous surface EMG and intramuscular EMG measurements will be acquired from the spastic biceps of the patients. Patients will be seated comfortably on a height-adjustable chair. The arm to be tested will be secured firmly on a customized apparatus with the elbow joint at approximately 90° of flexion and the shoulder at approximately 45° of abduction and 30° of flexion. The 128-channel unipolar surface EMG signals will be recorded with 2 flexible 2-dimensional 64-channel surface electrode array. A coating fine wire electrode will be inserted into the mid-axial section of the biceps to record bipolar intramuscular EMG signals. Ultrasound scan will be performed on the biceps to identify the location of the inserted wire electrode. Patients will be asked to contract their impaired biceps to perform maximum voluntary contraction of elbow flexion against the vertical plates 3 times.
  Arms: 3-dimensional innervation zone (3DIZ) guided injection

SUMMARY:
The purpose of this study is to evaluate if it is possible to use a new 3D imaging method to guide Botulinum neurotoxin (BTX) injection for muscle spasticity management after stroke. This imaging method is called three dimensional innervation zone imaging, or 3DIZI.

ELIGIBILITY:
Inclusion Criteria:

* a history of not more than one stroke which occurred at least 6 months prior to study enrollment;
* elbow flexor spasticity rated at 2 or 3 on Modified Ashworth scale (MAS);
* receiving repeated botulinum toxin injection every 3-4 months;
* absence of excessive pain in the paretic upper limb;
* capacity to provide informed consent, with Mini-Mental State Examination (MMSE) must be 25 or higher;

The following modified Ashworth scale (MAS) will be used for spasticity assessment:

0 -No increase in muscle tone; 1 -Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension; 1+ -Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM; 2 -More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved; 3 -Considerable increase in muscle tone, passive movement difficult; 4 -Affected part(s) rigid in flexion or extension.

Exclusion Criteria:

* recent botulinum toxin injection < 4 months;
* recent changes in antispastic medications <3 weeks (i.e., the antispastic medication regime is not stable;
* Changes in antispastic medications (such as baclofen, tizanidine, dantrolene etc) during the followup research visits. (NOTE: it is clinically rare for patients who receive repeated injections to change their antispastic medications);
* history of spinal cord injury or traumatic brain damage;
* history of serious medical illness such as cardiovascular or pulmonary complications;
* any condition that, in the judgment of a physician, would prevent the person from participating.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheng Li, MD, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard BTX Injection (Ultrasound Guided) | 3-dimensional Innervation Zone (3DIZ) Guided Injection
Started | 8 | 9
Completed | 7 | 8
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard BTX Injection (Ultrasound Guided) | 3-dimensional Innervation Zone (3DIZ) Guided Injection | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.43 (11.91) | 52.75 (11.90) | 54.00 (11.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 4 | 5 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1 | 0 | 1
  Black | 4 | 2 | 6
  Hispanic | 1 | 3 | 4
  Asian | 1 | 2 | 3
  Other | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Spasticity as Assessed by Reflex Torque of Elbow Flexors
Description: Each subject will receive a total of 60 degrees of computer-controlled elbow extension stretching at different speeds. The stretch ends at 10 degrees beyond the resting angle of the elbow joint during standing to offset the baseline difference among subjects. From the angle-torque relations, reflex torque is obtained after subtracting passive torque at 5˚/sec from those at 50˚/sec or 100˚/sec. Reflex torque is considered to reflect the neural component of muscle spasticity.
Time Frame: baseline (1 day prior to BTX injection)
Population: Data for 1 in each arm was not analyzed because these participants only completed one out of three sessions.
Measure: Mean (Standard Deviation); unit: Newton meter (n-m)
Arm/Group | Standard BTX Injection (Ultrasound Guided) | 3-dimensional Innervation Zone (3DIZ) Guided Injection
Number analyzed (Participants) | 7 | 8
Newton meter (n-m)
  reflex torque at 50˚/sec | 2.32 (1.73) | 2.04 (1.19)
  reflex torque 100˚/sec | 2.41 (2.35) | 3.11 (1.67)

2. Primary Outcome: Spasticity as Assessed by Reflex Torque of Elbow Flexors
Description: as for outcome 1
Time Frame: 3 weeks after BTX injection
Population: Data for 1 in each arm was not analyzed because these participants only completed one out of three sessions.
Measure: Mean (Standard Deviation); unit: Newton meter (n-m)
Arm/Group | Standard BTX Injection (Ultrasound Guided) | 3-dimensional Innervation Zone (3DIZ) Guided Injection
Number analyzed (Participants) | 7 | 8
Newton meter (n-m)
  reflex torque at 50˚/sec | 2.22 (1.21) | 1.47 (0.63)
  reflex torque at 100˚/sec | 2.64 (1.69) | 2.14 (1.20)

3. Primary Outcome: Spasticity as Assessed by Reflex Torque of Elbow Flexors
Description: as for outcome 1
Time Frame: 3 months after BTX injection
Population: Data for 1 in each arm was not analyzed because these participants only completed one out of three sessions.
Measure: Mean (Standard Deviation); unit: Newton meter (n-m)
Arm/Group | Standard BTX Injection (Ultrasound Guided) | 3-dimensional Innervation Zone (3DIZ) Guided Injection
Number analyzed (Participants) | 7 | 8
Newton meter (n-m)
  reflex torque at 50˚/sec | 2.71 (2.12) | 1.89 (0.75)
  reflex torque at 100˚/sec | 3.29 (2.57) | 2.85 (1.23)

4. Secondary Outcome: Spasticity as Assessed by the Modified Ashworth Scale (MAS)
Description: The following modified Ashworth scale (MAS) will be used for spasticity assessment:
  0 -No increase in muscle tone;
  1 -Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension;
  1+ -Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM; 2 -More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved; 3 -Considerable increase in muscle tone, passive movement difficult; 4 -Affected part(s) rigid in flexion or extension.
Time Frame: baseline (1 day prior to BTX injection)
Population: Data for 1 in each arm was not analyzed because these participants only completed one out of three sessions.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard BTX Injection (Ultrasound Guided) | 3-dimensional Innervation Zone (3DIZ) Guided Injection
Number analyzed (Participants) | 7 | 8
Participants
  0 | 0 | 0
  1 | 0 | 0
  1+ | 0 | 0
  2 | 7 | 6
  3 | 0 | 2
  4 | 0 | 0

5. Secondary Outcome: Spasticity as Assessed by the Modified Ashworth Scale (MAS)
Description: as for outcome 4
Time Frame: 3 weeks after BTX injection
Population: Data for 1 in each arm was not analyzed because these participants only completed one out of three sessions.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard BTX Injection (Ultrasound Guided) | 3-dimensional Innervation Zone (3DIZ) Guided Injection
Number analyzed (Participants) | 7 | 8
Participants
  0 | 0 | 0
  1 | 0 | 1
  1+ | 4 | 4
  2 | 3 | 2
  3 | 0 | 1
  4 | 0 | 0

6. Secondary Outcome: Spasticity as Assessed by the Modified Ashworth Scale (MAS)
Description: as for outcome 4
Time Frame: 3 months after BTX injection
Population: Data for 1 in each arm was not analyzed because these participants only completed one out of three sessions.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard BTX Injection (Ultrasound Guided) | 3-dimensional Innervation Zone (3DIZ) Guided Injection
Number analyzed (Participants) | 7 | 8
Participants
  0 | 0 | 0
  1 | 0 | 0
  1+ | 2 | 2
  2 | 5 | 5
  3 | 0 | 1
  4 | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Standard BTX Injection (Ultrasound Guided) | 3-dimensional Innervation Zone (3DIZ) Guided Injection
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 0/7 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-21): https://cdn.clinicaltrials.gov/large-docs/41/NCT03302741/Prot_SAP_000.pdf